CLINICAL TRIAL: NCT05637710
Title: Multicenter,Randomized,Parallel,Double-blind,Double-dummy,Comparative Superiority Study of Levocetirizine 5mg / Pseudoephedrine 240mg From Eurofarma vs Zina®5mg in the Symptomatic of Allergic Rhinitis
Brief Title: Parallel, Double-dummy, Superiority Study Levocetirizine/Pseudoephedrine x Zina for Allergic Rhinitis in Brazil
Acronym: ALERZIN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic change in development priorities
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EF180
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Participants who meet all eligibility criteria will be randomized to one of the following treatment groups:
  Investigational group: FDC levocetirizine 5mg / pseudoephedrine 240mg from Eurofarma Laboratórios S.A. (investigational drug) Participants randomized to this group will receive one (01) film-coated tablet of the investigational drug + one (01) levocetirizine placebo tablet, once a day, for seven (07) days.
  Comparator group: Levocetirizine 5mg (Zina® - comparator drug) Participants randomized to this group will receive one (01) levocetirizine 5mg tablet (Zina® 5mg) + one (01) FDC placebo tablet, once daily, for seven (07) days.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Investigational group: FDC levocetirizine 5mg / pseudoephedrine 240mg from Eurofarma Laboratórios S.A.
  Interventions: Drug: Administration of investigation of Eurofarma drug
- Group 2 (Active Comparator): Comparator group: Levocetirizine 5mg (Zina® - comparator drug)
  Interventions: Drug: Administration of Comparator

INTERVENTIONS:
Drug: Administration of investigation of Eurofarma drug — Participants randomized to this group will receive one (01) film-coated tablet of the investigational drug + one (01) levocetirizine placebo tablet, once a day, for seven (07) days.
  Other Names: Investigation drug
  Arms: Group 1
Drug: Administration of Comparator — Participants randomized to this group will receive one (01) levocetirizine 5mg tablet (Zina® 5mg) + one (01) FDC placebo tablet, once daily, for seven (07) days.
  Other Names: Comparator drug
  Arms: Group 2

SUMMARY:
AR is the most common respiratory disease worldwide and is clinically defined by the presence of nasal symptoms induced by exposure to allergens, particularly nasal obstruction and pruritus, runny nose and sneezing. The treatment purpose is to prevent or alleviate symptoms as safely and effectively as possible. Above all, it is recommended that patients avoid contact with allergens to which they are sensitive. However, this is often not enough, and pharmacological interventions are often required.

H1 antihistamines (anti-H1) are considered first-line drugs in the treatment of AR1. These drugs effectively relieve symptoms of the immediate phase of AR, such as nasal pruritus, sneezing, runny nose and associated eye symptoms, and partially the nasal blockage characteristic of the late phase of the disease. Due to their excellent safety profile and therapeutic advantages in the treatment of AR, second-generation anti-H1 drugs, such as levocetirizine, should always be prioritized over older compounds in all age groups1.

The combined administration of an antihistamine and an oral decongestant was shown to b more effective than the administration of an antihistamine alone for the relief of AR-associated nasal obstruction1.

Levocetirizine is an active pharmaceutical ingredient (API) registered in the country as a monodrug for oral administration at a dose of 5mg. Pseudoephedrine is not marketed as a monodrug for oral use in our area, but it is registered in FDC with antihistamines, which is why there is no comparator arm treating with pseudoephedrine only. These products are widely used and their efficacy and safety are well known in daily clinical practice in the proposed indication.

Once the absence of a pharmacokinetic interaction between levocetirizine and pseudoephedrine has been confirmed in relative bioavailability studies (RBA), this phase 3 study will be conducted in order to demonstrate the superiority of FDC levocetirizine 5mg / pseudoephedrine 240mg over levocetirizine 5mg administered alone in the symptomatic treatment of AR, particularly with regard to nasal obstruction. The registration seeks to provide a new effective and safe therapeutic option to address these cases.

DETAILED DESCRIPTION:
The investigational drug consists of a fixed-dose combination (FDC) that contains levocetirizine, a second-generation anti-H1 antihistamine agent, and pseudoephedrine, an oral decongestant, in doses of 5mg and 240mg, respectively, in the dosage form of film-coated tablets. This product is an unprecedented FDC in the country that is indicated for the symptomatic treatment of allergic rhinitis (AR) in patients aged ≥ 12 years.

A multicenter, randomized, parallel-group, double-blind, double-dummy, superiority, active-controlled clinical trial.

Adolescents and adults (aged ≥ 12 years) of both sexes with intermittent or persistent AR will be randomized in a 1:1 ratio to receive the investigational drug (FDC levocetirizine 5mg / pseudoephedrine 240mg from Eurofarma Laboratórios S.A.) or levocetirizine 5mg (Zina®), once daily (morning), for seven (07) days.

The severity of nasal allergy symptoms in the last 24 hours (nasal obstruction, runny nose, sneezing and nasal pruritus) will be evaluated through the application of the assessment questionnaire for nasal symptoms in the last 24 hours before, during and at the end of treatment. The severity of the nasal obstruction at that timepoint will also be evaluated immediately before and one (01) hour after the administration of the first dose of the study treatment, carried out at the research site (also in the morning). Participants will be monitored for an additional seven (07) days for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes who meet all of the following criteria will be enrolled in the study:

1. Signature of the Informed Consent Form (ICF) for those over 18 years of age and, when applicable, signature of the Informed Assent Form (IAF) by the participant under 18 years of age and the ICF by the legal representative before any study procedure.
2. Age ≥ 12 years and ≤ 65 years and weight ≥ 40 kg.
3. Clinical diagnosis of intermittent or persistent allergic rhinitis according to the definition of the Allergic Rhinitis and its Impact on Asthma2 (ARIA) group (Attachment 1) for at least two (02) years.

Exclusion Criteria:

Patients who meet at least one of the following criteria will be excluded from the study:

1. Concomitant presence of other types of rhinitis (such as infectious rhinitis, drug rhinitis, rhinitis in the elderly, hormonal rhinitis, non-allergic occupational rhinitis) when known.
2. Presence of significant septal deviation, compatible with impaired nasal ventilatory function, at the discretion of the investigator.
3. Presence of nasal polyposis on anterior rhinoscopy.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | In the last 24 hours determined seven (07) days after the ingestion of the first dose
  Absolute variation of the nasal obstruction score in the last 24 hours (VEON24D7) determined seven (07) days after the ingestion of the first dose of the IP in relation to the baseline score (VEON24D7 = EON24D7 - EON24D0), and the nasal obstruction scores correspond to the severity of this symptom in the last 24 hours (question 1 of the assessment questionnaire for nasal symptoms in the last 24 hours) and are evaluated on a 4-point categorical scale (0 = absent, 1 = mild, 2 = moderate and 3 = severe).

SECONDARY OUTCOMES:
Secondary efficacy endpoints | Absolute variation of the nasal obstruction score at that timepoint determined one (01) hour after the ingestion of the first dose
  • Absolute variation of the nasal obstruction score at that timepoint (VEONm1h) determined one (01) hour after the ingestion of the first dose of the IP in relation to the baseline score (VEONm1h = NEOm1h - NEOm0h), and the nasal obstruction scores at that timepoint correspond to the severity of this symptom at the time of evaluation and are evaluated on a 4-point categorical scale (0 = absent, 1 = mild, 2 = moderate and 3 = severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No